CLINICAL TRIAL: NCT04139135
Title: A Randomized, Double-blinded, Multicenter, Phase III Clinical Study of HLX10 (Recombinant Humanized Anti-PD-1 Monoclonal Antibody Injection) Combined With Chemotherapy Versus Placebo Combined With Chemotherapy for Neoadjuvant/Adjuvant Treatment of Gastric Cancer
Brief Title: A Clinical Study of HLX10 Combined With Chemotherapy Versus Placebo Combined With Chemotherapy for Neoadjuvant/Adjuvant Treatment of Gastric Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HLX10-006-GCneo
Record Dates: First submitted 2019-10-16; First posted 2019-10-25 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2022-06

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HLX10 (Experimental): HLX10 combined with chemotherapy will be adopted in the neoadjuvant treatment phase, and HLX10 monotherapy will be administered in the adjuvant treatment phase
  Interventions: Drug: HLX10
- Placebo (Placebo Comparator): Placebo combined with chemotherapy will be given in the neoadjuvant treatment phase, and chemotherapy alone will be administered during the adjuvant treatment phase.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: HLX10 — neoadjuvant treatment phase：HLX10（4.5mg/kg/3w IV） +SOX, adjuvant treatment phase：HLX10（4.5mg/kg/3w IV）
  Other Names: Recombinant humanized anti-PD-1 monoclonal antibody injection
  Arms: HLX10
Drug: Placebos — neoadjuvant treatment phase：placebos（4.5mg/kg/3w IV） +SOX, adjuvant treatment phase：SOX
  Arms: Placebo

SUMMARY:
This is a two-arm, randomized, double-blinded, multicenter phase III clinical study to evaluate the efficacy of HLX10 combined with chemotherapy versus placebo combined with chemotherapy for neoadjuvant/adjuvant treatment of gastric cancer.

Subjects will be randomized to the following two arms at 1: 1 ratio:

* Arm A (HLX10 arm): HLX10 combined with chemotherapy will be adopted in the neoadjuvant treatment phase, and HLX10 monotherapy will be administered in the adjuvant treatment phase;
* Arm B (control arm): Placebo combined with chemotherapy will be given in the neoadjuvant treatment phase, and chemotherapy alone will be administered during the adjuvant treatment phase.

Chemotherapy regimen SOX (oxaliplatin + tegafor gimeracil oteracil potassium (S-1)) will be used in the neoadjuvant treatment phase in Arm A and B, and in the adjuvant treatment phase in Arm B.

After randomization, subjects will receive a total of 3 cycles of neoadjuvant treatment with the mentioned treatment regimen.Surgery will be performed within 3-6 weeks after the last cycle of neoadjuvant treatment.All subjects who have completed the surgery will be unblinded after surgery, and adjuvant treatment will be started 3 to 12 weeks after surgery. Subjects randomized to Arm A (HLX10 arm) will continue to receive HLX10 monotherapy for up to 17 cycles (12 months).Subjects in Arm B after surgery (control arm) will continue to use chemotherapy alone (oxaliplatin + S-1) for 5 cycles.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary participation in the clinical study; fully understands and is informed of the study and has signed the Informed Consent Form (ICF); willing to comply with and able to complete all trial procedures.
2. The gender is not limited. When ICF is signed, the age is ≥ 18 years and ≤ 70 years old.
3. Histologically confirmed untreated gastric cancers, mainly adenocarcinoma.
4. Within 4 weeks prior to first dose, determined by the Independent Radiology Review Committee (IRRC) as: ≥ T3 and number of lymph node metastases ≥ 1 and no distant metastasis.
5. Prior to enrollment, the attending physician will evaluate to determine the eligibility for a R0 resection for the purpose of radical treatment.
6. Have good cardiac function and can be treated with radical resection.
7. tumor specimen testing results are PD-L1 positive (CPS ≥5). Subjects must provide the tumor tissues at screening or in the investigated surgery (if any), for PD-L1 expression level assessment.
8. Within 7 days before the first use of the study drug, ECOG: 0 ~ 1;
9. Expected survival 12 weeks;
10. The functions of the vital organs meet requirements.

Exclusion Criteria:

1. Existence of other active malignant tumors within 5 years or at the same time.
2. Plan to perform or have undergone an organ or bone marrow transplant.
3. Myocardial infarction and poorly controlled arrhythmias occurred within 6 months prior to the first dose.
4. Existence of grade III - IV cardiac disorders defined by the NYHA or echocardiogram shows: LVEF (left ventricular ejection fraction) < 50%.
5. Human immunodeficiency virus (HIV) infection.
6. Patients with active tuberculosis.
7. Patient with previous or current interstitial pneumonia, pneumoconiosis, radiation pneumonitis, drug-associated pneumonia, severely impaired lung function, etc.
8. Patients who have previously received other antibody/drug treatments for immune checkpoints, such as PD-1, PD-L1, and CTLA4 treatments.
9. Have diseases that may increase the risk of participating in the study and using the study medications, or other severe, acute, and chronic diseases and therefore are judged by the investigator to be unsuitable for clinical studies.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 642 (Estimated)
Dates: Start 2019-12-12 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
EFS | from randomizationuntil firstly confirmed and recorded disease progression or death (whichever occurs earlier),assessed up to 3 years
  event-free survival (assessed by independent radiological review committee (IRRC) based on RECIST v1.1)

SECONDARY OUTCOMES:
EFS | from randomizationuntil firstly confirmed and recorded disease progression or death (whichever occurs earlier)，assessed up to 3 years
  Event-free survival (assessed by the investigator per RECIST v1.1 criteria)
DFS | from the start of surgery to disease recurrence or death (for any reason)，assessed up to 3 years
  Disease-free survival (assessed by the investigator per RECIST v1.1 criteria)
pCR rate | after surgery，an average of 6 months
  Pathological complete response (pCR) rate (assessed by central pathology laboratory and the site)
5-year OS rate | OS is the time from randomization to death (of any cause)，assessed up to 5 years
  5-year overall survival (OS) rate

CONTACTS AND LOCATIONS:
Locations (15):
- China (15):
  - Peking University shenzhen hospital, Shenzhen, Guangdong
  - Affiliated Hospital of Hebei University, Baoding
  - Beijing Cancer Hospital, Beijing
  - China PLA General Hospital, Beijing
  - Peking University International Hospital, Beijing
  - Peking University Third Hospital, Beijing
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu
  - Cangzhou People's Hospital, Cangzhou
  - Anhui Provincial Hospital, Hefei
  - The First Affiliated Hospital of Anhui Medical University, Hefei
  - Linyi Cancer Hospital, Linyi
  - The Fourth Hospital of Hebei Medical University, Shijia Zhuang
  - Shanxi Provincial People's Hospital, Taiyuan
  - Tianjin Medical University Institute & Hospital, Tianjin
  - Xingtai People's Hospital, Xingtai